CLINICAL TRIAL: NCT01457690
Title: Study of the Absorption of Vitamin E Water-soluble Form (Pegylated) in the Familial Hypocholesterolemia With Chylomicron Retention
Acronym: VEDROP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010.634
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2015-11

CONDITIONS: Hypobetalipoproteinemias
Keywords: Vitamin E pegylated; chylomicron retention; Familial Hypocholesterolemia; Hypobetalipoproteinemias
MeSH Terms: conditions — Hypobetalipoproteinemias | interventions — tocophersolan; alpha-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tocofersolan: Vitamin E water-soluble (Experimental): 2 months off the conventional treatment before the study. Administration of a daily dose of vitamin E for 4 months
  Interventions: Drug: Tocofersolan
- Tocopherol alpha: Vitamin E conventional fat-soluble form (Active Comparator): 2 months off the conventional treatment before the study. Administration of a daily dose of vitamin E for 4 months
  Interventions: Drug: tocopherol alpha
- volunteers (Active Comparator)
  Interventions: Drug: Tocofersolan and tocopherol alpha

INTERVENTIONS:
Drug: Tocofersolan — Administration of a daily dose of vitamin E for 4 months:50 IU/kg
  Arms: Tocofersolan: Vitamin E water-soluble
Drug: tocopherol alpha — Administration of a daily dose of vitamin E for 4 months:50 IU/kg
  Arms: Tocopherol alpha: Vitamin E conventional fat-soluble form
Drug: Tocofersolan and tocopherol alpha — Administration of a single dose of vitamin E (Vitamin E water-soluble then Vitamin E conventional fat-soluble form)
  Arms: volunteers

SUMMARY:
To evaluate the kinetics of intestinal absorption of vitamin E water-soluble form from the classical lipid-soluble form in a population of patients with intestinal malabsorption (hypocholesterolemias family by retention of chylomicrons).

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from familial hypocholesterolemia by retention of chylomicrons
* Systematically followed in the department of Gastroenterology and Paediatric Nutrition in Women Mother Child's Hospital or in the endocrinology department of GHE (Louis Pradel Hospital);
* During treatment with oral vitamin E;
* over the age of 3 years and weighing over 16 kg at the time of inclusion
* For which there is a signed informed consent from the patient or parents / guardians in the case of a minor patient, and benefit from social security coverage.

Exclusion Criteria:

* Patient with encephalopathy
* Hypersensitivity to the active substance or the excipients of Vedrop
* A suspected allergy to local anaesthetics (including xylocaine)
* Patients who may not be compliant to treatment (psychiatric);
* In case of refusal to participate in the study from the patient and / or parents or legal guardian;
* Patients unable to consent (if patients with encephalopathy)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measurement the area under the curve of absorption of vitamin E according to its dosage form (fat-soluble versus water-soluble) in the beginning of each treatment period. versus water-soluble) in the beginning of each treatment period. | 12 months

SECONDARY OUTCOMES:
Measurement of serum (membranes erythrocytic) of vitamin E at the beginning and after each treatment. | 12 months
  Measurement of serum (membranes erythrocytic) of vitamin E at the beginning and after each treatment. Search for a correlation between the rates in adipose tissue and those in the membrane of erythrocytes.
Measurement of tissue (subcutaneous adipose tissue) of vitamin E at the beginning and after each treatment. | 12 months
  Measurement of tissue (subcutaneous adipose tissue) of vitamin E at the beginning and after each treatment. Search for a correlation between the rates in adipose tissue and those in the membrane of erythrocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Noel PERETTI, MD, PhD, Principal Investigator — Hopital Femme Mere Enfant, Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mere Enfant-Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Result] Cuerq C, Henin E, Restier L, Blond E, Drai J, Marcais C, Di Filippo M, Laveille C, Michalski MC, Poinsot P, Caussy C, Sassolas A, Moulin P, Reboul E, Charriere S, Levy E, Lachaux A, Peretti N. Efficacy of two vitamin E formulations in patients with abetalipoproteinemia and chylomicron retention disease. J Lipid Res. 2018 Sep;59(9):1640-1648. doi: 10.1194/jlr.M085043. Epub 2018 Jul 18. PMID 30021760